CLINICAL TRIAL: NCT06146829
Title: Development of Interpretable Machine Learning Models for Prediction of Acute Kidney Injury After Noncardiac Surgery
Brief Title: Machine Learning Models for Prediction of Acute Kidney Injury After Noncardiac Surgery
Status: Completed | Type: Observational
Sponsor: Rao Sun (Other)
Responsible Party: Sponsor-Investigator, Rao Sun, Associate chief physician, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJH-20230608C
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Acute kidney injury (AKI) is a common surgical complication characterized by a rapid decline in renal function. Patients with AKI are at an increased risk of developing chronic kidney disease and end-stage renal disease, which has been associated with an increased risk of morbidity, mortality and financial burdens. Identifying high-risk patients for postoperative AKI early can facilitate the development of preventive and therapeutic management strategies, and prediction models can be helpful in this regard.

The goal of this retrospective study is to develop prediction models for postoperative AKI in noncardiac surgery using machine learning algorithms, and to simplify the models by including only preoperative variables or only important predictors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) who had a serum creatinine measurement within 10 days before surgery and at least one measurement within 7 days after surgery.
* Eligible surgeries encompassed general, thoracic, orthopedic, obstetric, gynecology, and neurosurgery procedures lasting longer than 1 hour

Exclusion Criteria:

* Patients with concurrent cardiac, vascular, urological, or transplant surgeries.
* Patients with an American Society of Anesthesiologists (ASA) physical status V.
* Patients with end-stage renal disease (i.e., a glomerular filtration rate [eGFR] of 15 mL/min/1.73 m² or receiving hemodialysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent noncardiac surgical procedures at Tongji hospital between July 2018 and October 2022 were included.
Sampling Method: Non-Probability Sample
Enrollment: 88367 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Within 7 days after surgery
  In accordance with the KDIGO creatinine criteria: a serum creatinine increases of 26.5 mmol/L within 48 hours or 1.5 times baseline within 7 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rao Sun, Principal Investigator — Tongji Hospital
Locations (1):
- Rao Sun, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun R, Li S, Wei Y, Hu L, Xu Q, Zhan G, Yan X, He Y, Wang Y, Li X, Luo A, Zhou Z. Development of interpretable machine learning models for prediction of acute kidney injury after noncardiac surgery: a retrospective cohort study. Int J Surg. 2024 May 1;110(5):2950-2962. doi: 10.1097/JS9.0000000000001237. PMID 38445452